CLINICAL TRIAL: NCT00005236
Title: Atherosclerosis and Omega-3 Fatty Acids in Alaskan Natives
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1117; R01HL042082 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Artery Disease

SUMMARY:
To determine whether there were differences in the prevalence and extent of atherosclerotic lesions in the coronaries and aortas between Alaskan natives and non-natives, and whether the extent of the lesions was related to omega-3 fatty acids in blood and tissues.

DETAILED DESCRIPTION:
BACKGROUND:

Purported low mortality from coronary heart disease in Eskimos from Greenland, Canada, or Alaska has been interpreted by many investigators as synonymous with the absence of or reduced amount of atherosclerotic lesions in the coronary arteries compared to populations with a high rate of coronary heart disease. It was thought that this study would help to clarify the role of omega-3 fatty acids in atherosclerosis but also would help in making a decision whether to recommend to the general public the inclusion of fish oils, which contain large amounts of these fatty acids in the diet, for prevention and/or reduction of atherosclerotic heart disease.

DESIGN NARRATIVE:

Coronary arteries, aortas, blood, adipose tissue, and liver were collected at autopsy from deceased Alaskan natives, aged 5 years and above, dying of all causes and from a similar number of age- and sex-matched non-native Alaskans. Tested standardized methods of gross evaluation, histomorphometry, and chemistry were used to characterize, measure, and evaluate the prevalence and extent of atherosclerosis in arteries. Chemical methods for determination of blood and tissue lipids and gas liquid chromatographic methods for determination of fatty acids in various lipid fractions in plasma and tissues were used. Risk factors for coronary artery disease were evaluated from tissues taken at autopsy. Hypertension was evaluated by an examination of kidney arterioles. Cigarette smoking was evaluated by measurement of thiocyanate in the blood and the presence or absence of diabetes was evaluated by measuring glycosylation of hemoglobin from red blood cells. Findings were compared with those studied in other populations such as Blacks and whites in New Orleans, and Japanese, Norwegians and nineteen other ethnic groups in the International Atherosclerosis Project.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-12; Study Completion 1994-11 (Actual)

REFERENCES:
- [Background] Newman WP 3rd, Middaugh JP, Guzman MA, Propst MT, Rogers DR. Comparison of atherosclerosis in alaska Natives and nonnatives. Arch Pathol Lab Med. 1997 Oct;121(10):1069-75. PMID 9341586
- [Background] Batzer MA, Arcot SS, Phinney JW, Alegria-Hartman M, Kass DH, Milligan SM, Kimpton C, Gill P, Hochmeister M, Ioannou PA, Herrera RJ, Boudreau DA, Scheer WD, Keats BJ, Deininger PL, Stoneking M. Genetic variation of recent Alu insertions in human populations. J Mol Evol. 1996 Jan;42(1):22-9. doi: 10.1007/BF00163207. PMID 8576959
- [Background] Scheer WD, Boudreau DA, Malcom GT, Middaugh JP. Apolipoprotein E and atherosclerosis in Alaska Natives. Atherosclerosis. 1995 Apr 24;114(2):197-202. doi: 10.1016/0021-9150(94)05483-y. PMID 7605388
- [Background] Batzer MA, Stoneking M, Alegria-Hartman M, Bazan H, Kass DH, Shaikh TH, Novick GE, Ioannou PA, Scheer WD, Herrera RJ, et al. African origin of human-specific polymorphic Alu insertions. Proc Natl Acad Sci U S A. 1994 Dec 6;91(25):12288-92. doi: 10.1073/pnas.91.25.12288. PMID 7991620
- [Background] Newman WP, Middaugh JP, Propst MT, Rogers DR. Atherosclerosis in Alaska Natives and non-natives. Lancet. 1993 Apr 24;341(8852):1056-7. doi: 10.1016/0140-6736(93)92413-n. PMID 8096960
- [Background] Mulvad G, Pedersen HS, Hansen JC, Dewailly E, Jul E, Pedersen M, Deguchi Y, Newman WP, Malcom GT, Tracy RE, Middaugh JP, Bjerregaard P. The Inuit diet. Fatty acids and antioxidants, their role in ischemic heart disease, and exposure to organochlorines and heavy metals. An international study. Arctic Med Res. 1996;55 Suppl 1:20-4. PMID 8871682
- [Background] Boudreau DA, Middaugh JP, Mulvad G, Pedersen HS, Hansen JC, Malcom GT, Newman WP 3rd. Project meeting report: atherosclerosis & omega 3 fatty acids in Arctic Natives. Arctic Med Res. 1996 Jan;55(1):27-31. No abstract available. PMID 8901165